CLINICAL TRIAL: NCT02988622
Title: 1550-nm Non Ablative Laser (Fraxel) Versus Ablative 10,600-nm Carbon Dioxide (CO2) Fractional Laser in the Treatment of Surgical and Traumatic Scars: A Comparison Study on Efficacy, Treatment Regimen, and Cost.
Brief Title: Comparison of Lasers in the Treatment of Scars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marta Hemmingson-Van Beek (Other)
Responsible Party: Sponsor-Investigator, Marta Hemmingson-Van Beek, Sponsor Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201509722
Record Dates: First submitted 2016-11-28; First posted 2016-12-09 (Estimated); Results first posted 2017-12-08 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-03

CONDITIONS: Scar
MeSH Terms: conditions — Cicatrix | interventions — Lasers, Gas

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes

ARMS (1):
- Scar treated with Fraxel and CO2 laser (Other): One half of scar is treated with Fraxel laser and the other half of scar is treated with CO2 laser.
  Interventions: Device: Fraxel Laser; Device: CO2 Laser

INTERVENTIONS:
Device: Fraxel Laser — One half of the scar is treated with Fraxel Laser
Device: CO2 Laser — One half of the scar is treated with CO2 Laser.

SUMMARY:
The purpose of this study is to compare the 1550-nm non-ablative Fraxel laser (referred to as Fraxel Laser in this application) to the ablative 10,600-nm carbon dioxide fractional laser (referred to as CO2 Laser in this application) to determine if one is superior to the other in improving the appearance of scars over a series of three treatments. In addition, the investigators hope to identify a more cost-effective method to improve the appearance of scars caused by surgery or trauma.

DETAILED DESCRIPTION:
This study will be accomplished through a controlled split-scar study design whereby half of the scar will be treated with the Fraxel Laser and the other half of the scar will be treated with the CO2 Laser. This study is a blinded, prospective comparative, split-scar study whereby 100 participants will be recruited, enrolled and followed for a period of 9 months. The study population will include male and female participants, age 18 and over with scars secondary to surgery or trauma on any part of the body. The study will recruit participants with light colored skin, Fitzpatrick Type I-IV, because colored skin has a significantly higher risk of keloid scarring. The scar must measure a minimum of 4 cm in length to accommodate for the split-scar treatment. The participants will undergo laser treatments on Visit 1, Visit 2 and Visit 3 and each visit will be 4 weeks apart. The participants will return for evaluation and follow-up 3 months and 6 months following the last laser treatment. At each visit, photographs will be taken using identical camera settings, lighting and participant positioning. Evaluation of the scars will be completed by the participants and by blinded dermatology physicians. Participants will use a complete visual analogue scale at each visit, the Patient and Observer Scar Assessment Scale (POSAS) and a satisfaction score.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older.
2. Fitzpatrick skin type I-IV.
3. Scars secondary to surgery or trauma.
4. Scar length minimum 4 cm in length.

Exclusion Criteria:

1. Scars less than 6 weeks old.
2. History of keloid scarring.
3. Use of isotretinoin currently or within 3 months of enrollment
4. Use of photosensitive medication currently or within 3 months of enrollment.
5. Pregnancy -

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pooja Chitogopeker, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Health Care, Department of Dermatology, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 100 patients were recruited from the University of Iowa, Hospitals and Clinics between June to August 2016.
Pre-assignment Details: The exclusion criteria included any scar less than 6 weeks old, a history of keloid scarring, use of isotretinoin or other photosensitizing medication at the time of the study or within the previous 3 months and if the patient was pregnant.
Groups:
- Scar is Treated With Fraxel Laser and CO2 Laser: Each patient received treatment with both lasers to separate halves of their scar.
  Fraxel Laser: One half of the scar is treated with Fraxel Laser
  CO2 Laser: One half of the scar is treated with CO2 Laser.
Period: Overall Study
Arm/Group | Scar is Treated With Fraxel Laser and CO2 Laser
Started | 100
Completed | 83
Not Completed | 17
Not completed — Lost to Follow-up | 17

BASELINE CHARACTERISTICS:
Groups:
- Scar is Treated With Fraxel Laser and CO2 Laser: Fraxel Laser: One half of the scar is treated with Fraxel Laser
  CO2 Laser: One half of the scar is treated with CO2 Laser.
Arm/Group | Scar is Treated With Fraxel Laser and CO2 Laser
Number analyzed (Participants) | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 97
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.8 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80
  Male | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 100
Scar age [Mean (Standard Deviation); unit: years] | 11.7 (13.7)
Scar length [Mean (Standard Deviation); unit: Centimeters] | 12.1 (9.1)

OUTCOME MEASURES:

1. Primary Outcome: Scar Pain
Description: Patient and Observer Scar Assessment Scale (POSAS). Minimum of 1 and maximum of 10 (higher score is equivalent to a worse outcome). These are patient recorded scores.
Time Frame: Baseline and 6 months
Population: Patients with available data at the 6-month time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Scar is Treated With Fraxel Laser: Each patient received treatment with both lasers to separate halves of their scar.
  Fraxel Laser: One half of the scar is treated with Fraxel Laser
- Scar Treated With CO2 Laser: Each patient received treatment with both lasers to separate halves of their scar.
  Fraxel Laser: One half of the scar is treated with CO2 Laser
Arm/Group | Scar is Treated With Fraxel Laser | Scar Treated With CO2 Laser
Number analyzed (Participants) | 100 | 100
units on a scale
  Baseline | 1.265 (0.938) | 1.181 (0.608)
  6 months: number analyzed (Participants) | 83 | 83
  6 months | 1.048 (0.215) | 1.084 (0.474)
Statistical Analysis 1: Comparison: Scar is Treated With Fraxel Laser vs Scar Treated With CO2 Laser; Test type: Superiority; p = 0.0492, t-test, 2 sided; Mean Difference (Net) = 0.1205, Standard Deviation 0.5499

2. Primary Outcome: Scar Itching
Description: as for outcome 1
Time Frame: Baseline and 6 months
Population: Patients with available data at the 6-month time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Scar is Treated With Fraxel Laser | Scar Treated With CO2 Laser
Number analyzed (Participants) | 100 | 100
units on a scale
  Baseline | 1.386 (0.853) | 1.337 (0.873)
  6 months: number analyzed (Participants) | 83 | 83
  6 months | 1.084 (0.568) | 1.277 (1.140)
Statistical Analysis 1: Comparison: Scar is Treated With Fraxel Laser vs Scar Treated With CO2 Laser; Test type: Superiority; p = 0.0817, t-test, 2 sided; Mean Difference (Net) = 0.2410, Standard Deviation 0.0817

3. Primary Outcome: Scar Color
Description: as for outcome 1
Time Frame: Baseline and 6 months
Population: Patients with available data at the 6-month time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Scar is Treated With Fraxel Laser | Scar Treated With CO2 Laser
Number analyzed (Participants) | 100 | 100
units on a scale
  Baseline | 5.622 (2.623) | 5.518 (2.661)
  6 months: number analyzed (Participants) | 83 | 83
  6 months | 4.108 (2.078) | 4.313 (2.112)
Statistical Analysis 1: Comparison: Scar is Treated With Fraxel Laser vs Scar Treated With CO2 Laser; Test type: Superiority; p = 0.0686, t-test, 2 sided; Mean Difference (Net) = 0.3659, Standard Deviation 1.7951

4. Primary Outcome: Scar Stiffness
Description: as for outcome 1
Time Frame: Baseline and 6 months
Population: Patients with available data at the 6-month time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Scar is Treated With Fraxel Laser | Scar Treated With CO2 Laser
Number analyzed (Participants) | 100 | 100
units on a scale
  Baseline | 4.361 (2.770) | 4.518 (2.856)
  6 months: number analyzed (Participants) | 83 | 83
  6 months | 3.313 (2.112) | 3.386 (2.094)
Statistical Analysis 1: Comparison: Scar is Treated With Fraxel Laser vs Scar Treated With CO2 Laser; Test type: Superiority; p = 0.6278, t-test, 2 sided; Mean Difference (Net) = -0.0843, Standard Deviation 1.5789

5. Primary Outcome: Scar Thickness
Description: as for outcome 1
Time Frame: Baseline and 6 months
Population: Patients with available data at the 6-month time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Scar is Treated With Fraxel Laser | Scar Treated With CO2 Laser
Number analyzed (Participants) | 100 | 100
units on a scale
  Baseline | 5.325 (2.785) | 5.145 (2.833)
  6 months: number analyzed (Participants) | 83 | 83
  6 months | 3.373 (1.943) | 3.530 (2.086)
Statistical Analysis 1: Comparison: Scar is Treated With Fraxel Laser vs Scar Treated With CO2 Laser; Test type: Superiority; p = 0.0848, t-test, 2 sided; Mean Difference (Net) = 0.3373, Standard Deviation 1.7619

6. Primary Outcome: Scar Irregularity
Description: as for outcome 1
Time Frame: Baseline and 6 months
Population: Patients with available data at the 6-month time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Scar is Treated With Fraxel Laser | Scar Treated With CO2 Laser
Number analyzed (Participants) | 100 | 100
units on a scale
  Baseline | 6.602 (2.888) | 6.500 (2.616)
  6 months: number analyzed (Participants) | 83 | 83
  6 months | 3.3964 (2.167) | 4.084 (2.199)
Statistical Analysis 1: Comparison: Scar is Treated With Fraxel Laser vs Scar Treated With CO2 Laser; Test type: Superiority; p = 0.3418, t-test, 2 sided; Mean Difference (Net) = 0.2195, Standard Deviation 2.0788

7. Primary Outcome: Overall Opinion
Description: as for outcome 1
Time Frame: Baseline and 6 months
Population: Patients with available data at the 6-month time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Scar is Treated With Fraxel Laser | Scar Treated With CO2 Laser
Number analyzed (Participants) | 100 | 100
units on a scale
  Baseline | 6.695 (2.215) | 6.654 (2.265)
  6 months: number analyzed (Participants) | 83 | 83
  6 months | 4.024 (2.049) | 4.207 (2.187)
Statistical Analysis 1: Comparison: Scar is Treated With Fraxel Laser vs Scar Treated With CO2 Laser; Test type: Superiority; p = 0.1752, t-test, 2 sided; Mean Difference (Net) = 0.2375, Standard Deviation 1.5528

8. Primary Outcome: Patient Satisfaction
Description: Patients rated how satisfied they were with the appearance of each half of the treated scar.
Time Frame: 6 months
Population: Participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Scar is Treated With Fraxel Laser | Scar Treated With CO2 Laser
Number analyzed (Participants) | 83 | 83
Participants
  Very dissatisfied | 0 | 0
  Dissatisfied | 2 | 3
  Somewhat dissatisfied | 10 | 9
  Somewhat satisfied | 18 | 23
  Satisfied | 33 | 28
  Very Satisfied | 19 | 19
  Missing | 1 | 1

9. Primary Outcome: Observer Total Score
Description: Change in total observer score made up of components rating the scar appearance based on photos at baseline and photos at 6 months. Scale includes the following components: Visual analog scale from 0 to 10 (with 0 being excellent appearance and 10 being worst appearance), scar color, contour and distortion (these 3 measures were graded from 1 to 4 with 1 equating to perfect and 4 equating to worst appearance), scar finish (matte scar was given a score of 1 and shiny scar was given a score of 2). The total score of the above components provided an overall observer score, with 4 being the best score possible (equating to best appearing scar) and 24 being the worst score possible (equating to worst appearing scar).
Time Frame: Baseline and 6 months.
Population: Patients with available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Scar is Treated With Fraxel Laser | Scar Treated With CO2 Laser
Number analyzed (Participants) | 83 | 83
units on a scale | -0.3238 (1.9781) | 0.0586 (2.0552)
Statistical Analysis 1: Comparison: Scar is Treated With Fraxel Laser vs Scar Treated With CO2 Laser; Test type: Superiority; p = 0.0281, t-test, 2 sided; Mean Difference (Net) = 0.3824, Standard Deviation 1.5685

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Scar is Treated With Fraxel Laser | Scar Treated With CO2 Laser
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/100
Other Adverse Events (participants affected / at risk) | 3/100 | 3/100
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Scar is Treated With Fraxel Laser (N=100) | Scar Treated With CO2 Laser (N=100)
Blistering (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3) — Superficial blisters on the skin following treatment with CO2 and Fraxel laser

LIMITATIONS AND CAVEATS:
This is the largest split scar study comparing the C02 laser and Fraxel laser, however despite this the numbers are still relatively small overall. 100 patients were enrolled in teh study but only 83 completed the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-04-18): https://cdn.clinicaltrials.gov/large-docs/22/NCT02988622/SAP_000.pdf
  • Study Protocol (2017-11-16): https://cdn.clinicaltrials.gov/large-docs/22/NCT02988622/Prot_001.pdf